CLINICAL TRIAL: NCT06649383
Title: Virtual Reality for Elderly Patients in Anesthesia and Surgical Care
Brief Title: Virtual Reality (VR) Could Be a Good Alternative to Relaxing or Pain-relieving Medication
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pether Jildenstal (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Pether Jildenstal, Professor Pether Jildenstal Gothenburg University, Göteborg University
Organization: Göteborg University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-04059-01
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Virtual Reality; Distraction; Elderly (people Aged 65 or More)
Keywords: virtual reality; distraction

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR group (Experimental): This group use VR glasses during surgery
  Interventions: Device: Virtual reality
- Control group (No Intervention): Control group without intervention, conventional treatment

INTERVENTIONS:
Device: Virtual reality — Participant will try virtual reality glasses with tailormade software films to see if it's possible to use them as distraction during awake surgery. We will measure doses of propofol given, level of anxiety, experience of the patient and surgeons satisfaction.
  Arms: VR group

SUMMARY:
We want to investigate whether Virtual Reality (VR) could be a good alternative to the relaxing or pain-relieving medications that are often used to alleviate anxiety when patients undergo surgery under local anesthesia.

DETAILED DESCRIPTION:
This study is a randomized controlled trial based on both quantitative and qualitative methods. Inclusion criteria are elderly patients aged ≥65 years with an estimated surgery time of a maximum of 90 minutes, who undergo surgery/treatment under local anesthesia and sedation. Randomization is to either standard sedation or sedation/VR. Randomization is carried out using mixed, sealed envelopes. The studies will be conducted at the following locations:

Hallands Hospital, Kungsbacka: Open inguinal hernia surgery with implant, anesthesia type is infiltration anesthesia.

Sahlgrenska Hospital: Intervention, cannulation of the groin and vascular surgery performed via catheters/guides on blood vessels, liver, pancreas, and abdominal organs, with anesthesia type infiltration.

Alingsås Hospital: Surgery on the hand, arm, lower extremity, urology, with anesthesia type block and infiltration.

Data collection will include baseline preoperative stress levels measured with The State-Trait Anxiety Inventory (STAI-S) and pain assessment using a numerical rating scale (NRS) from 0-11.

We also plan to use an objective marker for measuring anxiety-induced stress perioperatively, such as heart rate variability or skin conductance measurement. Postoperative data will include STAI-S, NRS, intraoperative sedative medication (type and dosage in mg/kg), time to urination, time to oral nutrition, discharge time, and time spent in the postoperative ward.

The patient will assess their well-being with the QoR 15 and NRS during the first five days postoperatively. The patient will be contacted to schedule a follow-up individual interview with semi-structured questions via Zoom two weeks after the surgery.

The primary outcome effect of VR glasses on mg/kg of propofol used intraoperatively or another sedative drug and/or the amount of local anesthetic used in mg. The secondary outcome effect of VR glasses on anxiety-induced stress perioperatively, where data collection will be conducted using EEG spectral edge frequency and The State-Trait Anxiety Inventory (STAI-S).

ELIGIBILITY:
Inclusion Criteria:

* over 65 years, planed surgery in local anesthesia/regional anesthesia

Exclusion Criteria:

* dementia, unable to cooperate, cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2029-06-15 (Estimated)

PRIMARY OUTCOMES:
propofol mg/kg | during the surgery (90 minutes max)
  dose of propofol given during surgery to the participant

SECONDARY OUTCOMES:
Surgeons satisfaction | Directly after surgery is finished
  surgeons satisfaction, measured with NASA task load index (tlx). Higher score, worse outcome.
Stress/anxiety | during the surgery (90 minutes max)
  Stress or anxiety felt during surgery by participant, measured with State-Trait Anxiety Inventory (STAI) . Higher score worse outcome.
Nurse anesthetists experience, (questionnaire). | Directly after surgery is finished
  Nurse anesthetists experience will be measured with a questionnaire egarding how well the monitoring of the patient could be carried out and the degree to which the patient was perceived as calm. The higher score, the better.
Level of pain | Directly after surgery is finished
  Patients level of pain after surgery, measured with Numeric rating scale (NRS). The higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Alingsås lasarett, Alingsås, Västra Götaland County
  - Sahlgrenska universitetssjukhuset, Gothenburg, Västra Götaland County

IPD SHARING:
Plan to Share IPD: No